CLINICAL TRIAL: NCT02566018
Title: Treatment Options for Proximal Humerus Fractures in the Elderly and Their Implication on Personal Independence
Brief Title: Treatment of Proximal Humerus Fractures in the Elderly
Acronym: prox_hum
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-310
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Humeral Fractures
Keywords: elderly
MeSH Terms: conditions — Humeral Fractures | interventions — Therapeutics; Equipment and Supplies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- experimental intervention: A greater degree of initial displacement is tolerated to allow for conservative, non-operative treatment in more simple fracture patterns. Two-part fractures with marked displacement including two part patterns with a non-displaced greater or minor tuberosity fracture (formally three part fractures) are treated with a proximal humerus nail; and displaced three and four part fractures are primarily managed with a reverse total shoulder arthroplasty. Proximal Humeral Internal Locking System (PHILOS)-plates are only used exceptionally in this group of patients.
  Interventions: Procedure: treatment/medical device
- control intervention: Since May 2013 we have changed our treatment algorithm for the treatment of fractures of the humeral head in the elderly. Before this change in algorithm we used PHILOS plates extensively and rarely Inverse Shoulder prostheses.
  In general all proximal humerus fractures were operated except minimally or undisplaced.
  Interventions: Procedure: standard

INTERVENTIONS:
Procedure: treatment/medical device — The new treatment algorithm was applied to all patients with proximal humerus fracture as from May 2013 onwards
  Groups: experimental intervention
Procedure: standard — The old treatment algorithm was applied to all patients with proximal humerus fracture up to May 2013.
  Groups: control intervention

SUMMARY:
This study is set to evaluate a proposed standard for the treatment of proximal humerus fractures

DETAILED DESCRIPTION:
This study investigates the effect of routine treatment algorithm for proximal humerus fractures. All applied treatments are approved and reflect routine practice. The follow-up investigation as planned for this study is associated with only minimal risk for the concerned patients.

ELIGIBILITY:
Inclusion Criteria:

* Age of 65 years or above
* Proximal humerus fracture
* Informed consent by the patient or legal representatives to participate in the study

Exclusion Criteria:

* More than one fracture, polytrauma
* Suspicion of a pathological fracture in the context of known or unknown malignancy
* Previous surgery of the proximal humerus on the same side
* High energy trauma
* Open Fracture
* Insufficient German language skills

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients fulfilling all of the following inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
personal dependency status | 6 months
  A simple four point rating is used at the time of injury (for the premorbid state) and at 6 months to demonstrate the impact of the injury (including its treatment) on the ability to return to the former social environment and degree of self-dependency.

SECONDARY OUTCOMES:
range of motion | 6 months
Shoulder pain and disability index (SPADI) | 6 months
  The SPADI is a patient-based questionnaire containing 15 questions about pain and activities of daily living that must be answered by the patient on a scale of 0-10 (0 = no pain / no difficulties to 10 = Worst pain / activity). Five questions relate to the pain and 8 questions relate to the function in daily activities, both subscores are combined and converted to the total score to 0 (= lowest score) to 100 (= best result). A validated German version is available
SSV | 6 months
  The Subjective Shoulder Value (SSV) is based on a single question that is answered subjectively by the patients. The English formulation of this question is: "What is the overall percent value of your shoulder if a completely normal shoulder represents 100%?" 12 It is an easily administered measure of shoulder function.
General health using EuroQuality of life (EQ)-5D-5L visual analogue scale (VAS) | 6 months
  The gain in quality of life within two years after surgery is assessed using the generic Quality of Life (QoL) EuroQoL EQ-5D-5L instrument.
Quality of life (utilities) derived using EQ-5D-5L | 6 months
  Using the EQ-5D-5L instrument patients are asked to report on their general health status on a VAS scale from 0 (worst possible health) to 100 (best possible health).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rikli, Prof, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Result] Schurch MA, Rizzoli R, Mermillod B, Vasey H, Michel JP, Bonjour JP. A prospective study on socioeconomic aspects of fracture of the proximal femur. J Bone Miner Res. 1996 Dec;11(12):1935-42. doi: 10.1002/jbmr.5650111215. PMID 8970896
- [Result] Rikli D, Feissli S, Muller AM, Steinitz A, Suhm N, Jakob M, Audige L. High rate of maintaining self-dependence and low complication rate with a new treatment algorithm for proximal humeral fractures in the elderly population. J Shoulder Elbow Surg. 2020 Jun;29(6):1127-1135. doi: 10.1016/j.jse.2019.11.006. Epub 2020 Feb 10. PMID 32057657